CLINICAL TRIAL: NCT05375617
Title: Southern European Prospective Investigation Into Childhood Cancer and Nutrition (EPICkids)
Brief Title: European Prospective Investigation Into Childhood Cancer
Acronym: EPICkids
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: AAAU1164
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; Brain Tumor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Brain Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute lymphoblastic leukemia cohort
  Interventions: Other: Observational
- Brain tumor cohort
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention

SUMMARY:
Over the last decades, research has shown that poor nutritional status can adversely impact prognosis and increase toxicities during treatment for childhood cancer. EPICkids is a collaboration between the International Initiative for Pediatrics and Nutrition, the International Agency for Research on Cancer, and sites throughout three Southern European countries (Spain, Greece, and Italy). The primary aim of EPICkids is to establish an informational resource on critical nutrition parameters wherein we can describe the trajectory of nutritional status among Southern European children and adolescents with acute lymphoblastic leukemia (ALL) and favorable biology brain tumors, investigate lifestyle behaviors, sociodemographic factors, and quality of life and correlate these indicators with clinical outcomes. The specimens obtained with the proposed study will foster future studies on nutrition and prevalent childhood cancer as well as establish a framework to develop evidence-based guidelines for European children with cancer, utilizing regional, European data. We plan to recruit 900 patients with ALL and 1400 patients with a favorable biology brain tumor over five years. Nutrition parameters and lifestyle factors will be measured at systematic timepoints over the study period. Stool and blood specimens will be collected at each timepoint. Eligible patients will be between 3 and 21 years of age.

DETAILED DESCRIPTION:
Over the last decades, research has shown that poor nutritional status can adversely impact prognosis and increase toxicities during treatment for childhood cancer. EPICkids is a collaboration between the International Initiative for Pediatrics and Nutrition, the International Agency for Research on Cancer, and sites throughout three Southern European countries (Spain, Greece, and Italy). The primary aim of EPICkids is to establish an informational resource on critical nutrition parameters wherein we can describe the trajectory of nutritional status among Southern European children and adolescents with acute lymphoblastic leukemia (ALL) and favorable biology brain tumors, investigate lifestyle behaviors, sociodemographic factors, and quality of life and correlate these indicators with clinical outcomes. We will also create a prospective biorepository of specimens (stool, blood) obtained at diagnosis, during treatment, at the end of treatment, and after treatment among children and adolescents undergoing treatment for ALL and favorable biology brain tumors. We plan to recruit 900 patients with ALL and 1400 patients with a favorable biology brain tumor over five years. Eligible patients will be between 3 and 21 years of age receiving standard treatment at one of the participating institutions. Data will be collected at systematic timepoints over the study period and include demographics, food security, clinical data and disease characteristics, quality of life, physical activity, dietary intake, and nutritional anthropometric data. Blood and stool specimens will be collected at each timepoint throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

Age: ALL and favorable biology brain tumors: Patient must be between 3 years and 21 years of age at the time of consent.

Diagnosis:

* ALL: Patients must have newly diagnosed B-cell ALL, T-cell ALL, or mixed phenotype acute leukemia confirmed by immunophenotyping by flow cytometry.
* Brain tumors: Patients must have newly diagnosed favorable biology brain tumor confirmed by either pathology report, imaging and/or biochemical studies including low-grade gliomas, medulloblastoma, ependymoma, pituitary tumors, germ cell tumors.

Treatment:

* ALL and brain tumors: Participants may be children on a clinical trial or "as per" a clinical trial.
* ALL: Patients will receive standard leukemia treatment.
* Brain tumors: Patients will be treated depending upon standard approach with surgery, chemotherapy, radiation therapy. Patients receiving autologous stem cell transplantation as part of their regimen may be included.

Location: ALL and brain tumors: Patients must be receiving treatment at one of the participating centers.

Timing:

* ALL: Parents/guardians must consent and patient assent, if applicable, within three working days of diagnosis.
* Brain tumors: Parents/guardians must consent and assent, if applicable, prior to initiation of chemotherapy, radiation or stem cell transplant.

Exclusion Criteria:

ALL and brain tumors:

* Patients with relapsed or progressive disease, exclusive of patients with unresectable low-grade gliomas who have progressive disease.
* Patients with history of other primary malignancy.
* Patients with other medical conditions not associated with the malignancy that may interfere with nutritional status/growth and/or microbiome composition, like patients with Down's syndrome, metabolic disorders or celiac disease. Patients with genetic predisposition that may interfere with nutritional status/growth.

ALL:

* Patient plans to receive hematopoietic stem cell transplant.
* Mixed lineage leukemias who receive AML-based protocols. Brain tumors: Children/adolescents who will be managed by observation or surgery only, or diagnosed with ATRT or high-grade gliomas.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Southern European children and adolescents ages 3-21 years of age with acute lymphoblastic leukemia and favorable biology brain tumors.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the association of dietary and lifestyle variables to examine the association of nutritional status and dietary intake with side-effects from treatment and survival in children and adolescents with ALL and favorable biology brain tumors. | From diagnosis to 1 year post-end of treatment

SECONDARY OUTCOMES:
Examine the association of nutritional status and quality of life in children and adolescents with ALL and favorable biology brain tumors. | From diagnosis to 1 year post-end of treatment
Develop evidence-based, regional guidelines on dietary intake and nutritional status in children and adolescents diagnosed with ALL and favorable biology brain tumors. | From diagnosis to 1 year post-end of treatment
Provide evidence-based, regional guidelines in order to standardize the delivery of nutritional care during and after cancer treatment for children and adolescents with ALL and favorable biology brain tumors. | From diagnosis to 1 year post-end of treatment
Create a prospective biorepository of specimens (stool, blood) obtained at diagnosis, during treatment, at the end of treatment, and after treatment among children and adolescents undergoing treatment for ALL and favorable biology brain tumors. | From diagnosis to 1 year post-end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elena J Ladas, PhD, RD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perganti F, Huybrechts I, Balduzzi AC, Barr R, Biondi A, Blade AL, Munoz Bravo E, Damasco E, Katsagoni CN, Kattamis A, Lassaletta A, Llopis Lera M, Llort A, Blanco Lopez J, Perez Martinez A, Massimino M, Morales La Madrid A, Moreno L, Munoz Alonso A, Nicolas G, Preziati G, Rizzari S, Della Valle S, Marquez Vega C, Walters M, Kozlakidis Z, Ladas EJ. Southern European Prospective Investigation Into Childhood Cancer and Nutrition (EPICkids): Study design and protocol. PLoS One. 2025 Sep 5;20(9):e0319110. doi: 10.1371/journal.pone.0319110. eCollection 2025. PMID 40911561